CLINICAL TRIAL: NCT00256100
Title: Assessment of the Safety and Efficacy of Fondaparinux as an Anticoagulant in Haemofiltration in Patients With Acute Renal Failure.
Brief Title: Fondaparinux as an Anticoagulant in Haemofiltration in Patients With Acute Kidney Failure.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Teh Priincipal investigator responsible for the trial no longer employed at the study site.
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004.066
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-04

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One (Active Comparator): Enoxaparin Sodium (Clexane ) is to be used in the control arm of the study
  Interventions: Drug: Fondaparinux Sodium
- Two (Active Comparator): Fondaparinux will be used as the anticoagulant in the sencond arm of the study
  Interventions: Drug: Fondaparinux Sodium

INTERVENTIONS:
Drug: Fondaparinux Sodium — The active group of the study will be given fondaparinux 10mg/24 hours for haemofiltration anticoagulation
  Other Names: Arixtra

SUMMARY:
The purpose of this project is to assess the safety and effectiveness of fondaparinux, a new drug to prevent blood clotting in the continuous dialysis machine used in intensive care patients who have kidney failure.

DETAILED DESCRIPTION:
The study hypothesis is that when used as an anticoagulant in haemofiltration, fondaparinux prolongs the filter life when compared to enoxaparin.

Fondaparinux is the first compound of a new class of synthetic oligosaccharides with antithrombotic effects. It represents the active portion of the natural heparin molecule.

The null hypothesis is that there is no difference in filter life when using fondaparinux or enoxaparin as anticoagulation for haemofiltration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years or over) admitted to the ICU and expected to stay for more than 48 hours.
2. Patients who require continuous renal replacement therapy.
3. Patients who consent or if the patient is not competent, the next of kin who consent to inclusion in the study. .

   -

Exclusion Criteria:

1. Patients aged less than 18 years of age.
2. Patients who are pregnant
3. Patients with a contraindication to anticoagulation for pre existing bleeding diathesis
4. Patients or next of kin who do not consent to study inclusion. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The study will evaluate the duration of filter patency using fondaparinux as an anticoagulant in haemofiltration and compare this to the current standard haemofilter anticoagulant, enoxaparin. | Duration of the haemofilter life

SECONDARY OUTCOMES:
To assess the incidence of complications, primary bleeding with fondaparinux compared to enoxaparin in this setting. | Until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: John F Cade, Principal Investigator — Melbourne Health
Locations (1):
- The Royal Melbourne Hospital Intensive Care Unit Grattan Street, Parkville, Victoria, Australia